CLINICAL TRIAL: NCT00003726
Title: A Phase I/II Study of Recombinant Desulfato Hirudin, Lepirudin (Refludan) in Small Cell Lung Cancer Patients Previously Treated With Chemotherapy
Brief Title: Lepirudin in Treating Patients With Recurrent or Advanced Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study funding was dropped.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9815; P30CA023108 (NIH); DMS-9815 (Other: Dartmouth-Hitchcock Medical Center); NCI-V98-1512 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-05-03 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — lepirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lepirudin (Experimental): Dose level 1: 10 mg once daily -> (total dose, 10 mg/d) Dose level 2: 15 mg once daily -> (total dose, 15 mg/d) Dose level 3: 10 mg twice daily -> (total dose, 20 mg/d) Dose level 4: 15 mg twice daily -> (total dose, 30 mg/d) Dose level 5. 20 mg twice daily -> (total dose, 40 mg/d) Dose level 6: 25 mg twice daily -> (total dose, 50 mg/d)
  Interventions: Biological: lepirudin

INTERVENTIONS:
Biological: lepirudin — lepirudin

SUMMARY:
RATIONALE: Anticoagulants, such as lepirudin, may help prevent blood clots from forming in patients who have received chemotherapy for small cell lung cancer.

PURPOSE: This phase I/II trial is studying the side effects and best dose of lepirudin in treating patients with recurrent or advanced small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the dose, safety, and antitumor response rate of lepirudin in patients with recurrent or extensive stage small cell lung cancer previously treated with chemotherapy.

OUTLINE: This is a dose escalation (in individual patients) study. Patients receive dose escalated lepirudin subcutaneously once or twice a day for 3-4 days. Dose escalation continues in each patient until aPTT prolongation occurs or the maximum dose level is reached. The patient then continues treatment on the maximum tolerated dose. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 20-35 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

1. Pathologically confirmed recurrent or extensive stage small cell lung cancer.
2. Received at least one prior chemotherapy regimen
3. Measurable or evaluable disease that has not been irradiated
4. No pleural effusions, bone metastases, brain metastases, elevated serum enzymes, or radionuclide scans as the sole indicator lesion
5. Brain metastases allowed if patients received cranial irradiation and have no clinical evidence of brain metastases

PATIENT CHARACTERISTICS:

1. Age: Not specified
2. Performance status: Karnofsky 60-100%
3. Life expectancy: Not specified
4. Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3
5. Hepatic: Bilirubin no greater than 2.0 mg/dL PT and aPTT normal
6. Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min
7. Cardiovascular: No unstable heart rhythm No unstable angina No clinical evidence of congestive heart failure No prior cerebrovascular accident or stroke No uncontrolled or severe hypertension
8. Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception
9. At least 6 weeks since any signs or symptoms of bleeding No history of bleeding disorder
10. No bacterial endocarditis or other active infection

PRIOR CONCURRENT THERAPY:

1. Biologic therapy: Not specified
2. Chemotherapy: At least 3 weeks since prior chemotherapy
3. Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy
4. Surgery: At least 6 weeks since major surgery, trauma, or needle biopsy of any organ
5. Other: No concurrent anticoagulant or platelet inhibitor therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 1998-11; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R. Rigas, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was enrolled to the trial and started on 10mg and increased to 20mg. However developed progression of disease and was removed from the trial.
Pre-assignment Details: Funding was pulled and therefore the trial was not completed.
Period: Overall Study
Arm/Group | Lepirudin
Started | 1
Completed | 0 (Funding was pulled on the trial and therefore no other participants were enrolled)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lepirudin
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose, Safety and Antitumor Response Rate of Administering Recombinant Desulfato Hirudin, Elpirudin to Previously Treated Patients With Extensive or Recurrent Small Cell Lung Cancer
Description: Evaluated through clinical exams, tumor assessments, laboratory assessment, and adverse event assessments.
Time Frame: 18 months
Population: No data were collected
Arm/Group | Lepirudin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Lepirudin
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The funding of the trial was discontinued and therefore only one participant was enrolled to the trial and experienced no adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No